CLINICAL TRIAL: NCT02369120
Title: The Influence of a Biopsychosocial Educational Internet-based Intervention on Pain, Dysfunction, Quality of Life, and Pain Cognition in Chronic Low Back Pain Patients in Primary Care: a Mixed Methods Approach
Brief Title: Influence of a Educational Internet-based Intervention in Chronic Low Back Pain Patients: A Mixed Methods Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Francesc Valenzuela Pascual, Principal investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULleida
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Low Back Pain
Keywords: patient education; pain cognitions
MeSH Terms: conditions — Low Back Pain | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Normal care by GP (Active Comparator): Control group: Will follow conventional treatment provided by the family physician in primary care. This treatment is based on the clinical guidelines of the "Institut Català de la Salut" (http://www.gencat.cat/ics/professionals/guies/docs/guia_lumbalgies.pdf).
  Interventions: Other: Normal care by GP
- Educational intervention using a website (Experimental): This group of subjects will be given access to our web-site in where they will find information related to CLBP. This information will be provided in different formats: explanatory video by the author, animated video about the neurophysiology of pain, written format using metaphors, and FAQs. All this information will be based on the information provided by the subjects on QUAL. The aim of this educational intervention is to change patient´s misbeliefs about CLBP with the last outcome of reducing pain intensity, improving function, and reducing disability.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — The internet platform will provide patients with customized tasks that allow them to use the metaphor of the journey (the narrative as a dynamic of the game) to feel that they manage their own path, which will change negative perceptions into positive perceptions about certain actions. At all times, the patients will be able to choose among different information sources, such as videos about the origin of chronic pain, 3D representations of different neurophysiological processes, and FAQs. Additionally, the patients will be able to contact a specialist in the neurophysiology of pain by email or videoconference. Furthermore, to reinforce patients' motivation and participation, gamification techniques will be implemented.
  Arms: Educational intervention using a website
Other: Normal care by GP — Patients will follow GP advice including NSAID medication if needed
  Arms: Normal care by GP

SUMMARY:
Aim: The aim of this project is to identify chronic low back pain patients´ beliefs about the origin and meaning of pain for developing a biopsychosocial web-based educational intervention. The other aim of this project is to assess the effectiveness of this web-based educational intervention for chronic low back pain patients on pain cognitions, pain intensity, and disability.

Methods: Mixed methods design, combining both qualitative and quantitative methodologies. For the qualitative part of this study, the investigators will use qualitative in-depth semi-structured interviews. For the quantitative phase we will use an experimental study design.

Subjects: Chronic low back pain patients between 18-65 years old, attending a primary care setting in the city of Lleida.

Expected outcomes: The investigators expect to change and modify chronic low back pain patients´ cognition by using our web-site educational intervention, with the further outcome of reducing pain and disability.

DETAILED DESCRIPTION:
Hypothesis and outcomes

Hypothesis:

1. Persistent chronic low back pain and its consequences are maintained by the lack of understanding about the origin and meaning of pain.
2. Pain neurophysiology as an educational internet- based intervention for chronic low back pain will change cognition about the origin and meaning of pain, with the outcome of pain reduction, disability reduction, and better quality of life compared to normal care.

Outcomes:

There are specific objectives for each phase of the study.

Phase 1 (QUAL):

To identify chronic low back pain patients' beliefs concerning the origin and meaning of pain.

Phase 2 (Connecting procedure):

To construct and develop a biopsychosocial web- based educational intervention using the QUAL results.

Phase 2 (QUAN):

Primary outcome. To evaluate the effect of a biopsychosocial web-based educational intervention for chronic low back pain based on pain intensity compared to normal care.

Secondary outcomes. To assess the effect of a biopsychosocial web-based educational intervention for chronic low back pain compared to normal care on:

* Fear avoidance beliefs.
* Kinesiophobia.
* Disability.

Methodology Study design

To answer the research question, the authors will use a mixed-method sequential exploratory design. The pur- pose of mixed methodology is not to replace qualitative or quantitative methodologies, but to use the strengths of both while reducing their weaknesses. Specific- ally, the sequential exploratory design includes an initial qualitative phase followed by a quantitative phase, with the aim of developing an educational tool. In this project, we propose that both phases (qualitative and quantitative) must have the same relevance (QUAL- QUAN) for the development of the educational tool and that the development of the study must be conducted in three stages:

1. Qualitative data collection through semi-structured personal interviews followed by thematic analysis.
2. Construction of the educational tool with the results obtained in the previous step (topics or emerging categories).
3. Analysis of the effectiveness of the educational tool using a randomized controlled trial.

Scope: Primary care

SUBJECTS:

The recruitment process will be performed independently in each phase of the study, although in both phases this recruitment process will take place in the same pri- mary care centers in the city of Lleida through family physicians. The inclusion and exclusion criteria are also common to both phases. Prior to the beginning of the first phase, the first author of this study will perform a presentation of the project to the medical and nursing staff in each of the primary care centers involved in the study to ask for their cooperation.

QUAL: In this phase, patients will be recruited by their respective family physicians. Once the physician makes the diagnosis of CLBP and ensures that the individual meets the inclusion and exclusion criteria, the physician informs the patient about the existence of this project and invites him to contact the first author by telephone. If the person agrees to participate in the study, the inter- view will be scheduled to take place in the Faculty of Nursing and Physiotherapy of the University of Lleida.

QUAN: The recruitment process will start after the end of QUAL and the development of the educational tool. This phase will consist of an educational interven- tion using a randomized controlled trial design. The re- cruitment process will be the same as in QUAL. Prior to the beginning of the intervention, the first author will meet the study subjects individually to inform them of the study conditions and provide them with the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. History of CLBP longer than 6 months.
2. Patients between 20-65 years old.
3. To be able to read, speak and understand Spanish, Catalan, or English.
4. With access to the Internet, a computer or laptop and e-mail address.
5. To accept and sign the informed consent.

Exclusion Criteria:

* 1. Any red flag condition:

  * Onset age < 20 or > 55 years
  * Non-mechanical pain (unrelated to time or activity)
  * Thoracic pain
  * Previous history of carcinoma, steroids, HIV
  * Feeling unwell
  * Weight loss
  * Widespread neurological symptoms
  * Structural spinal deformity

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  This scale was developed by Huskinson in 1976 as a method of measuring pain intensity. VAS is an easy, simple and reproductible tool that can be used by the same patient in multiple occasions. The scale consists on a 10-cm line with a description on both extremes. In the far left "no pain", and "worst pain ever" in the far right of the scale. For some authors VAS is the most sensitive measure in clinical pain research
Fear Avoidance Beliefs | 2 weeks
  The FABQ is a self-reported questionnaire that consists of 16 items about the beliefs of LBP patients on the influence that physical activity and work have on their pain. Each item can be scored from 0 (totally agree) to 6 (totally disagree). The Spanish version of the FABQ has demonstrated good reliability
Kinesiophobia | 2 weeks
  This scale is widely used in pain medicine for assessing pain-related fear. The Spanish format has 11 items, with each scoring ranging from 1 (totally disagree) to 4 (totally agree). The Spanish version of the TSK is easy to use, reliable and valid

SECONDARY OUTCOMES:
Disability | 2 weeks
  This is a self-reported questionnaire assessing function and disability. It is an easy instrument for patients where scoring goes from 0 to 24, being clinically important a change of 4 or more points. RMQ is reliable, valid, and adequate to assess disability in patients with LBP. It has been successfully validated into Spanish

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Molina Luque, sociologist, Study Director — Universitat de Lleida; Rosa Gil Iranzo, Physics, Study Director — Universitat de Lleida; Francisco Corbi, Sports, Study Director — Universitat de Lleida; Jorge Soler Gonzalez, MD, Study Director — Universitat de Lleida
Locations (1):
- All Primary care settings, Lleida, Spain

REFERENCES:
- [Derived] Valenzuela-Pascual F, Molina F, Corbi F, Blanco-Blanco J, Gil RM, Soler-Gonzalez J. The influence of a biopsychosocial educational internet-based intervention on pain, dysfunction, quality of life, and pain cognition in chronic low back pain patients in primary care: a mixed methods approach. BMC Med Inform Decis Mak. 2015 Nov 23;15:97. doi: 10.1186/s12911-015-0220-0. PMID 26597937
- Available data/document: Study Protocol — http://www.biomedcentral.com/1472-6947/15/97